CLINICAL TRIAL: NCT01210469
Title: Effectiveness of Two Treatments on Posture and Balance in Elderly Women With Osteoporosis: a Randomized Clinical Trial
Brief Title: Effectiveness of Two Treatments on Posture and Balance in Elderly Women With Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Thomaz Nogueira Burke, Ms, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 787/06
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2008-03

CONDITIONS: Osteoporosis
Keywords: elderly; postural balance; musculoskeletal equilibrium; posture; muscle strength; muscle stretching exercises
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Strengthening Group (Experimental): Performed balance training with lower limbs muscle strengthening.
  Interventions: Other: Strengthening and balance exercises
- Stretching Group (Experimental): Performed balance training with stretching
  Interventions: Other: Stretching and balance exercises
- Control Group (No Intervention)

INTERVENTIONS:
Other: Strengthening and balance exercises — The group trained for 8 weeks, with sessions of about 60 minutes, twice a week.
  Other Names: Force Platform; Balance Master
  Arms: Strengthening Group
Other: Stretching and balance exercises — The group trained for 8 weeks, with sessions of about 60 minutes, twice a week.
  Other Names: Force Platform; Balance Master
  Arms: Stretching Group

SUMMARY:
The purpose of this study was compare the efficacy of two exercise programs - the first consisting of balance training and muscle strength and the second consisting of balance training and muscle stretching exercises - to improve postural control in elderly women with osteoporosis.

DETAILED DESCRIPTION:
The decrease in postural control and muscle strength in lower limbs have been identified as major risk factors for falls in older people. Exercises have proven effective in decreasing risk factors in healthy elderly, but little is known about the effects of interventions with exercise in the elderly with osteoporosis.

Objective: To compare the efficacy of two exercise programs - the first consisting of balance training and muscle strength and the second consisting of balance training and muscle stretching exercises - to improve postural control in elderly women with osteoporosis.

Methods: Fifty elderly aged 65 or older, with a diagnosis of osteoporosis, were randomized into 3 groups: Strength Group (n = 17) performed balance training with muscle strengthening; Stretching Group (n = 17) performed balance training with stretching; and Control Group (n =16) did not do activity. The groups trained for 8 weeks, with sessions of about 60 minutes, twice a week. Postural control was evaluated by Modified Clinical Test of Sensory Interaction for Balance (CTSIBm) and Limits of Stability test (LOS) in Balance Master force plate, the functional balance by Berg Balance Scale (BBS), muscle strength by dynamometry, the shortening of the hamstrings by goniometry and posture by PAS/SAPO (Postural Assessment Software).

ELIGIBILITY:
Inclusion Criteria:

* women from 65 to 80 yrs of age
* diagnosis of osteoporosis classified according to the criteria of the World Health Organization, with bone mineral densitometry reduced by at least 2.5 SD when compared with young adults (region of lumbar spine)

Exclusion Criteria:

* severe visual deficiency
* physically incapable of participating in the tests
* neurological disorders, amputations, or prostheses
* individuals with regular physical activity (twice or more per week) or who had recently participated in exercise programs for muscular strength or balance

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Postural Control | eight weeks
  Postural control was evaluated by Modified Clinical Test of Sensory Interaction for Balance (CTSIBm) and Limits of Stability test (LOS) in Balance Master force plate

SECONDARY OUTCOMES:
Postural alignment | eight weeks
  Postual alignment (thoracic kyphosis and forward head) measured by PAS/SAPO (Postural Assessment Software)
Lower limb muscle strength | eight weeks
  The muscle strength in knee extension and knee flexion was evaluated by dynamometry.
Shortening of the hamstrings | eight weeks
  The shortening of the hamstrings was evaluated by goniometry.
Berg Balance Scale | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomaz N Burke, MSc, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Link to my thesis in portuguese — http://www.teses.usp.br/teses/disponiveis/5/5163/tde-08032010-162215/